CLINICAL TRIAL: NCT07197177
Title: PECTORAL PLANE BLOCK COMPAIRED TO ERECTOR SPINAE PLANE BLOCK IN MULTIMODAL ANALGESIA FOR MASTECTOMY PATIENTS IN SOUTH ASIAN POPULATION -A PROSPECTIVE RANDOMISED CONTROL TRIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-21-22
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cancer
Keywords: Regional anesthesia
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PECTORAL PLANE BLOCK (Experimental): We will infiltrate local anesthesia in Pectoral Plane under ultrasound guidance.
  Interventions: Procedure: regional block
- ERECTOR SPINAE PLANE BLOCK (Experimental): We will infiltrate local anesthesia in ERECTOR spine Plane under ultrasound guidance.
  Interventions: Procedure: regional block

INTERVENTIONS:
Procedure: regional block — We will infiltrate local anesthesia (Bupivicaine 0.25 %), in pectoral plane vs Erecter spine plane, will observe intraoperative morphine consumption, pain scores and Pacu stay.

SUMMARY:
This prospective randomized controlled trial was conducted at the Department of Anesthesia, Shaukat Khanum Memorial Cancer Hospital and Research Centre (SKMCH&RC), Lahore. The sample size was calculated based on a previous study by Gad M. (2019) on patients undergoing modified radical mastectomy , where the mean morphine consumption in first 24 hours post operatively was reported as 16.7 ± 7.21 mg in the erector spinae plane (ESP) block group and 10.7 ± 3.12 mg in the pectoral plane block (PECS) group. Using the formula for comparison of two means with unequal standard deviations, and assuming a 90% power, 95% confidence interval, and a 10% dropout rate, the required sample size was determined to be 42 patients, with 21 patients in each group.

DETAILED DESCRIPTION:
This prospective randomized controlled trial was conducted at the Department of Anesthesia, Shaukat Khanum Memorial Cancer Hospital and Research Centre (SKMCH&RC), Lahore. The sample size was calculated based on a previous study by Gad M. (2019) on patients undergoing modified radical mastectomy , where the mean morphine consumption in first 24 hours post operatively was reported as 16.7 ± 7.21 mg in the erector spinae plane (ESP) block group and 10.7 ± 3.12 mg in the pectoral plane block (PECS) group. Using the formula for comparison of two means with unequal standard deviations, and assuming a 90% power, 95% confidence interval, and a 10% dropout rate, the required sample size was determined to be 42 patients, with 21 patients in each group

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status II or III, biopsy proven breast cancer, and were undergoing unilate l modified radical mastectomy

Exclusion Criteria:

* . Exclusion criteria included patient refusal to participate, age less than 18 years, diagnosed allergy or contraindication to local anesthetic, chronic pain, obesity (BMI >35), non-cancerous or undiagnosed breast lesions, ASA IV status, and emergency surgery.

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
Mean Morphine consumption | 12 hours
  calculate morphine consumption intraoperatively and post operative at 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Skmch & Rc, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided